CLINICAL TRIAL: NCT01260012
Title: Study on the Role of Antioxidant Micronutrients on the Reversal of Schistosomal Peri-portal Fibrosis of the Liver.
Brief Title: Antioxidant Supplements in the Reversal of Schistosomal Peri-portal Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Addis Ababa University (Other)
Collaborators: Ullevaal University Hospital (Other); University of Oslo (Other); University of Agder (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Dr Nega Berhe, Aklilu Lemma Institute of Pathobiology, Addis Ababa Ethiopia
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/794-1
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-09

CONDITIONS: Schistosomiasis; Liver Fibrosis; Periportal Fibrosis; Oxidative Stress
Keywords: Schistosoma mansoni; Schistosomiasis; periportal fibrosis; antioxidant; fibrosis reversal
MeSH Terms: conditions — Schistosomiasis; Liver Cirrhosis | interventions — Praziquantel; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- praziquantel+antioxidant (Experimental): Praziquantel therapy will be offered at the start, at six weeks and at 12 weeks from date of enrollment. Thereafter praziquantel therapy will be offered if subjects have demonstrable S. mansoni eggs on the subsequent six-monthly evaluations. In additions, antioxidant suppliment will be given daily for a period of one year
  Interventions: Dietary Supplement: Praziquantel+antioxidant suppl; Dietary Supplement: Praziquantel+antioxidant
- Praziquantel +placebo 2mths then antioxidant for 10 months (Active Comparator): Praziquantel therapy will be offered at the start, at six weeks and at 12 weeks from date of enrollment. Thereafter praziquantel therapy will be offered if subjects have demonstrable S. mansoni eggs on the subsequent six-monthly evaluations. In addition subjects will receive placebo as a supplement for two months which will be followed by antioxidant as a supplement for the rest of the year.
  Interventions: Other: Praziquantel + placebo 2mths then antioxidant for 10 mths
- Praziquantel therapy with placebo supplement (No Intervention): Praziquantel therapy will be offered at the start, at six weeks and at 12 weeks from date of enrollment. Thereafter praziquantel therapy will be offered if subjects have demonstrable S. mansoni eggs on the subsequent six-monthly evaluations. In addition subjects will receive placebo as a supplement for a period of one year.
  Interventions: Dietary Supplement: Praziquantel therapy and placebo as supplement

INTERVENTIONS:
Dietary Supplement: Praziquantel+antioxidant suppl — Praziquantel therapy will be offered at the start, at six weeks and at 12 weeks from date of enrollment. Thereafter praziquantel therapy will be offered if subjects have demonestrable S. mansoni eggs on the subsequent six-monthly evaluations. In addition subjects will receive antioxidant supplement on daily basis for a period of one year.
  Arms: praziquantel+antioxidant
Other: Praziquantel + placebo 2mths then antioxidant for 10 mths — Praziquantel therapy will be offered at the start, at six weeks and at 12 weeks from date of enrollment. Thereafter praziquantel therapy will be offered if subjects have demonestrable S. mansoni eggs on the subsequent six-monthly evaluations. In addition subjects will receive placebo as a supplement for two months which will be followed by antioxidant as a supplement for the rest of the year.
  Arms: Praziquantel +placebo 2mths then antioxidant for 10 months
Dietary Supplement: Praziquantel therapy and placebo as supplement — Praziquantel at day 0, 6-weeks and at 12 weeks from start of study. Thereafter praziquantel therapy will be offered if subjects have demonestrable s.mansoni eggs on six-monthly evaluation periods. Placebo will be given as a supplement for one year.
  Other Names: Placebo; Praziquantel
  Arms: Praziquantel therapy with placebo supplement
Dietary Supplement: Praziquantel+antioxidant — Praziquantel treatment will be offered at time 0, six weeks and 12 weeks from the start. Antioxidant supplement will be offered on a daily basis for a period of one year
  Other Names: Interventional
  Arms: praziquantel+antioxidant

SUMMARY:
Liver fibrosis is the most serious complication of schistosomiasis mansoni. However only limited proportion of subjects with infection develop this pathology and there is limited knowledge on risk factors for the differential morbidity patterns observed in endemic communities. Our preliminary cross-sectional study indicated that serum levels of antioxidants may be related with the development of fibrosis. The present project is a randomised double blinded placebo controlled prospective study investigating the role of food based antioxidant supplements on the outcome of anti-schistosomal chemotherapy with regards to the extent of fibrosis reversal.

DETAILED DESCRIPTION:
Schistosomiasis is the second leading parasitic disease worldwide, after malaria. Liver fibrosis is the most serious complication of schistosomiasis mansoni which can lead to reduced work capacity and early death in endemic countries. There is, however, limited knowledge on the development of liver fibrosis and the differential patterns morbidity observed in endemic communities. Our preliminary cross-sectional study in Ethiopia seems to indicate that serum levels of antioxidants may influence the development of fibrosis. The present project is a translational study combining basic antioxidant laboratory work with is a randomised double blinded placebo controlled prospective study in endemic areas in Ethiopia, investigating the role of food based antioxidant supplements on the outcome of anti-schistosomal chemotherapy with regards to the extent of fibrosis reversal. In addition, analysis of dietary intakes of antioxidants among communities with comparable levels of S. mansoni infection but with differing levels of schistosomal periportal fibrosis will be undertaken to compare serum levels of antioxidants and prevalence of liver fibrosis. Furthermore we plan to assess development of schistosomal peri-portal fibrosis in a cohort of students established 9 years back who had comparable levels of community prevalence of schistosomiasis but with differing access to fruits and vegetables. Research on this topic has a high priority globally which is in line with the millennium development goals. Knowledge in this field will also add to our understanding of fibrosis development in general and to the efficacy of clinical treatment of schistosomiasis in particular.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with schistosomal periportal fibrosis will be eligible for the study

Exclusion Criteria:

* Subjects with acute malaria, tuberculosis or other chronic diseases such as diabetes mellitus, cardiovascular disease or cancer will be excluded from the study.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 414 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Effect of antioxidant supplement on fibrosis reversal following praziquantel therapy | 2 years
  Patients schistosomal periportal fibrosis will be treated with praziquantel at the start, at six weeks and at 3 months from the start of the study. Praziquantel therapy will then be offered if subjects have demonstrable S. mansoni eggs on six-monthly evaluation periods. In addition, one group will recieve supplemental antioxidant for one year, the second group will recieve supplement as a placebo for two months and then antioxidant suppliment for 10 months, the third group will receive placebo as a supplement for one year.

SECONDARY OUTCOMES:
Time required for the reversal of schistosomal periportal fibrosis | 4 years
  Subjects will be followed with six-monthly evaluations for a period of 4 years and praziquantel therapy will be offered if subjects have demonstrable S. mansoni eggs on the six-monthly evaluations. Over the four year period we plan to assess the time required for the reversal of the various stages of schistosomal periportal fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Nega Berhe, MD, PhD, Principal Investigator — Aklilu Lemma Institute of Pathobiology, Addis Ababa University; Svein G Gundersen, MD PhD, Study Director — Sorlandet Hospital HF, Box 416, 4604 Kristiansand - Norway; Bjørn Myrvang, MD, PhD, Study Chair — Ullevål University Hospital, Department of Infectious Diseases, Centre for Imported and Tropical Diseases, 0407 Oslo; Rune Blomhoff, MSc, PhD, Principal Investigator — Institute for Basic Medical Sciences, Department of Nutrition, University of Oslo, P.O.box 1046, N-0316 Oslo, Norway
Locations (1):
- Aklilu Lemma Institute of Pathobiology, Addis Ababa University, Addis Ababa, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Berhe N, Halvorsen BL, Gundersen TE, Myrvang B, Gundersen SG, Blomhoff R. Reduced serum concentrations of retinol and alpha-tocopherol and high concentrations of hydroperoxides are associated with community levels of S. mansoni infection and schistosomal periportal fibrosis in Ethiopian school children. Am J Trop Med Hyg. 2007 May;76(5):943-9. PMID 17488920
- [Background] El-Sokkary GH, Omar HM, Hassanein AF, Cuzzocrea S, Reiter RJ. Melatonin reduces oxidative damage and increases survival of mice infected with Schistosoma mansoni. Free Radic Biol Med. 2002 Feb 15;32(4):319-32. doi: 10.1016/s0891-5849(01)00753-5. PMID 11841922
- [Background] Berhe N, Myrvang B, Gundersen SG. Reversibility of schistosomal periportal thickening/fibrosis after praziquantel therapy: a twenty-six month follow-up study in Ethiopia. Am J Trop Med Hyg. 2008 Feb;78(2):228-34. PMID 18256420
- [Background] Karlsen A, Paur I, Bohn SK, Sakhi AK, Borge GI, Serafini M, Erlund I, Laake P, Tonstad S, Blomhoff R. Bilberry juice modulates plasma concentration of NF-kappaB related inflammatory markers in subjects at increased risk of CVD. Eur J Nutr. 2010 Sep;49(6):345-55. doi: 10.1007/s00394-010-0092-0. Epub 2010 Feb 2. PMID 20119859
- [Background] Paur I, Austenaa LM, Blomhoff R. Extracts of dietary plants are efficient modulators of nuclear factor kappa B. Food Chem Toxicol. 2008 Apr;46(4):1288-97. doi: 10.1016/j.fct.2007.09.103. Epub 2007 Nov 5. PMID 17980947
- [Background] Blomhoff R. Dietary antioxidants and cardiovascular disease. Curr Opin Lipidol. 2005 Feb;16(1):47-54. doi: 10.1097/00041433-200502000-00009. PMID 15650563
- [Background] Eboumbou C, Steghens JP, Abdallahi OM, Mirghani A, Gallian P, van Kappel A, Qurashi A, Gharib B, De Reggi M. Circulating markers of oxidative stress and liver fibrosis in Sudanese subjects at risk of schistosomiasis and hepatitis. Acta Trop. 2005 May;94(2):99-106. doi: 10.1016/j.actatropica.2005.03.001. Epub 2005 Apr 7. PMID 15814296
- [Background] Halliwell B. The antioxidant paradox. Lancet. 2000 Apr 1;355(9210):1179-80. doi: 10.1016/S0140-6736(00)02075-4. No abstract available. PMID 10791396
- See also: Financial support for the research project was obtained from Ulleval hospital, Centre for Imported and Tropical Diseases — http://ulleval.no